CLINICAL TRIAL: NCT06503354
Title: Validation of Gait Metrics From Cionic Neural Sleeve
Brief Title: Gait Metric Validation of the Cionic Neural Sleeve
Status: Completed | Type: Observational
Sponsor: Cionic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB-FY2024-253
Record Dates: First submitted 2024-07-02; First posted 2024-07-16 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Validation Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Participants: Healthy adults
  Interventions: Device: Neural Sleeve and Zeno walkway

INTERVENTIONS:
Device: Neural Sleeve and Zeno walkway — A standard manual stopwatch will be used to record time. The Zeno pressure gait mat will be laid flat on the ground and used for all walking conditions/speed. Participants will perform two 5-minute walking bouts for each of the four walking conditions while wearing the Neural Sleeve without electrical stimulation. For normal walking speed, participants walked at their normal, comfortable pace for 5 minutes. For fast walking speed, participants walked to cover as much distance as possible for 5 minutes. For intermittent-slow speed, participants were instructed to walk as if browsing in a museum. For slow speed, participants walked at a slow, steady pace. The order of conditions was randomized. They will walk back and forth along a 12-meter course with the gait mat in the center of the course. Participants will not receive any intervention or treatment. Simultaneously, the Zeno walkway will be operated according to manufacturer's instructions.

SUMMARY:
The purpose of this study is to determine the validity of the Neural Sleeve gait metrics compared to gait parameters assessed with a Protokinetics Zeno pressure sensitive walkway. The spatiotemporal gait parameters obtained from the Zeno walkway have been rigorously validated and will represent the "gold standard" ground truth measurements in the proposed protocol. Confirming the validity of the Neural Sleeve metrics offers benefit to individuals who utilize the device by providing confidence that calculated gait reports are accurate and can be used to inform usage of the device and associated gait changes over time. Findings of inaccuracy would still offer benefit in the form of knowing that the Neural Sleeve metrics need to be used with caution and/or updated to provide correct outcomes to users.

DETAILED DESCRIPTION:
The study aims to validate the gait metrics of the Neural Sleeve in healthy adult volunteers. All participants will wear a Neural Sleeve on their dominant leg. The Zeno pressure gait mat will be laid flat on the ground and used for all four walking conditions. Participants will perform two 5-minute walking bouts at each of the four speed conditions while wearing the Cionic Neural Sleeve without electrical stimulation. The movement sensors on the Neural Sleeve will collect motion data that permits the comparison of gait metrics from the Neural Sleeve to those measured by the gait mat. During the walking trials, participants will be told that they can take a break if needed. Condition order will be randomized and participants will be offered 5 minutes of rest between consecutive trials. Validity of gait metrics of the Neural Sleeve will be compared against the Zeno walkway.

ELIGIBILITY:
Inclusion Criteria:

* Persons between the ages of 22-64
* Ability to ambulate at least 30 minutes during a two-hour period

Exclusion Criteria:

* Lower motor neuron disease or injury (e.g. peripheral neuropathy)
* Absent sensation in the legs
* Demand-type cardiac pacemaker or defibrillator
* Malignant tumor in the legs
* Existing thrombosis in the legs
* History of lower limb injury or orthopedic issues leading to impaired walking

Ages: 22 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2024-07-08 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-11 (Actual)

PRIMARY OUTCOMES:
Gait speed | A walking session of up to 5 minutes
  Time one takes to walk a specified distance (expressed as a ratio between distance and time, in centimeters per second)
Stride length | A walking session of up to 5 minutes
  Distance (centimeters) covered when one takes two steps, one with each foot, measured from ipsilateral heel contact to the next ipsilateral heel contact (right-to-right or left-to-left heel) (centimeters)
Cadence | A walking session of up to 5 minutes
  Number of steps per minute (steps per minute)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland State University, Department of Health Sciences and Human Performance, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No